CLINICAL TRIAL: NCT07147556
Title: Surgical Treatment of Functional Popliteal Artery Entrapment Syndrome: Results of a Systematic Approach Based on the Section of the Medial Gastrocnemius Attachment
Acronym: SAPP-F
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP251098; 2025-A01670-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Popliteal Artery Entrapment Syndrome
Keywords: Functional popliteal artery entrapment syndrome; Surgical treatment; Systematic approach; Athlete; Decompression
MeSH Terms: conditions — Popliteal Artery Entrapment Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Functional popliteal artery entrapment syndrome (FPAES) is a rare unique clinical entity that does not have associated with anatomic abnormalities and, therefore, is thought to be functional in nature (1,2). It has been first described by Rignault et al. in 1985, and its true mechanism is not well understood (3,4). Given the relative lack of knowledge of FPAES in the literature and the reported outcomes after decompressive surgery are limited and not standardized. The objective of this study was to describe our diagnostic and peri-operative protocol, clinical outcomes of a unique surgical management technique based on the systemic section of the attachment of the medial head of the gastrocnemius.

DETAILED DESCRIPTION:
This study is a single-center retrospective study of all patients who underwent surgical treatment of FPAES between 2015 and 2025 by 2 vascular surgeons. Patients will be identified via hospital database and data collection including patients' demographics, clinical presentation, length of hospitalisation, participation in sport, diagnostic workup, procedural details and complications, clinical improvement, and postoperative imaging were prospectively collected from a dedicated institutional database. To evaluate objectively the functional improvement as well as to assess the effectiveness of the surgical intervention, the Lower Extremity Functional Scale (LEFS) was used post operatively at the time of conducting this study. The LEFS is a self-administered questionnaire, comprised of 20 items, to assess patient's ability to perform everyday tasks and has been used by clinicians as a measure of patients' lower extremity initial function, ongoing progress and outcome after surgical intervention as well as to evaluate the functional impairment of lower extremities.

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent surgical treatment of functional popliteal artery entrapment syndrome between 2015 and 2025 and agree to participate in the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent surgical treatment of FPAES between 2015 and 2025
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical and functional improvement, and the return to the sportive level | at 1 year
  Clinical improvement was defined as the ability to increase activity or decreased discomfort of the initial presenting symptoms.
  To evaluate objectively the functional improvement as well as to assess the effectiveness of the surgical intervention, the Lower Extremity Functional Scale (LEFS) will be used post operatively at 1 year post operativeley

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël COSCAS, MD, PhD, Principal Investigator — CHU Ambroise Paré - APHP

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh N. Functional popliteal entrapment: A diagnostic and treatment conundrum. J Vasc Surg. 2019 Nov;70(5):1563. doi: 10.1016/j.jvs.2019.02.019. No abstract available. PMID 31653376
- [Background] Hislop M, Kennedy D, Cramp B, Dhupelia S. Functional Popliteal Artery Entrapment Syndrome: Poorly Understood and Frequently Missed? A Review of Clinical Features, Appropriate Investigations, and Treatment Options. J Sports Med (Hindawi Publ Corp). 2014;2014:105953. doi: 10.1155/2014/105953. Epub 2014 Sep 7. PMID 26464888
- [Background] Rignault DP, Pailler JL, Lunel F. The "functional" popliteal entrapment syndrome. Int Angiol. 1985 Jul-Sep;4(3):341-3. PMID 3831156
- [Background] Turnipseed WD. Functional popliteal artery entrapment syndrome: A poorly understood and often missed diagnosis that is frequently mistreated. J Vasc Surg. 2009 May;49(5):1189-95. doi: 10.1016/j.jvs.2008.12.005. PMID 19394547
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543